CLINICAL TRIAL: NCT07346755
Title: Effects of Suprascapular Nerve Block on Proprioception in Hemiplegic Shoulder Pain: A Randomized Controlled Trial
Brief Title: Suprascapular Nerve Block and Proprioception in Hemiplegic Shoulder Pain: A Randomized Controlled Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, merve kocibar, Medical Doctor, Fatih Sultan Mehmet Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SSNB-PT
Record Dates: First submitted 2026-01-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Hemiplegic Shoulder Pain; Proprioception; Suprascapular Nerve Block
Keywords: Hemiplegic Shoulder Pain; Proprioception; Suprascapular nerve block; Hemiplegia
MeSH Terms: conditions — Hemiplegia | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: A controlled, investigator-blinded, prospective parallel-group study.
Who Masked: Investigator
Masking Description: The study is planned as an investigators-blinded study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suprascapular Nerve Block (Experimental): Participants in this arm will receive a suprascapular nerve block administered by an experienced physician, followed by a standardized physical therapy and rehabilitation program. The nerve block will be performed using local anesthetic to reduce shoulder pain and facilitate participation in rehabilitation.
  Interventions: Procedure: suprascapular nerve block; Other: physical therapy
- Control (Active Comparator): Participants in this arm will receive a standardized physical therapy and rehabilitation program alone, without suprascapular nerve block. The program will be identical to that provided to the experimental arm and will follow routine clinical practice for hemiplegic shoulder pain.
  Interventions: Other: physical therapy

INTERVENTIONS:
Procedure: suprascapular nerve block — An ultrasound-guided suprascapular nerve block will be performed by injecting 5 mL of 2% lidocaine (Lidon 100 mg/5 mL solution for injection) into the suprascapular fossa.
  Arms: Suprascapular Nerve Block
Other: physical therapy — Accepted routine physical therapy modalities for hemiplegic shoulder pain, including cold pack application, transcutaneous electrical nerve stimulation, assisted shoulder range of motion exercises, and posterior capsule stretching exercises, will be administered five days per week for three weeks, in 45-minute sessions, for a total of 15 sessions

SUMMARY:
The purpose of this prospective randomized controlled clinical trial is to evaluate the effect of suprascapular nerve block on shoulder joint proprioception in stroke patients with hemiplegic shoulder pain.

Fourteen patients aged 18-80 years with hemiplegic shoulder pain will be randomized into two groups. One group will receive suprascapular nerve block followed by a standardized physical therapy program, while the control group will receive the same physical therapy program alone.

The primary outcome is shoulder joint proprioception. Secondary outcomes include pain intensity, shoulder range of motion, motor recovery, stroke-specific quality of life, and upper extremity functional outcomes.

The results of this study are expected to clarify the role of suprascapular nerve block on proprioception and rehabilitation outcomes in patients with hemiplegic shoulder pain.

DETAILED DESCRIPTION:
Hemiplegic shoulder pain is one of the most common painful complications following stroke, with a reported prevalence ranging from 16% to 84%. Its etiology is multifactorial and primarily includes musculoskeletal pathologies such as adhesive capsulitis, bicipital tendinitis, subacromial bursitis, shoulder subluxation, and rotator cuff disorders. Pain that may be present even at rest or during passive movement, along with reduced shoulder range of motion, represents the leading clinical complaint. Therefore, the main goal of treatment is to reduce pain, increase joint range of motion, and consequently enhance participation in rehabilitation and functional capacity.

Suprascapular nerve block is a widely used intervention to reduce pain and improve shoulder range of motion in patients with hemiplegic shoulder pain. Proprioceptive and nociceptive receptors embedded in the glenohumeral joint capsule and surrounding ligaments play a crucial role in joint stability, and the suprascapular nerve provides major innervation to these structures. Despite its widespread use to facilitate rehabilitation and improve outcomes, the effects of suprascapular nerve block on shoulder joint proprioception and the subsequent impact of potential proprioceptive changes on rehabilitation outcomes have not yet been investigated.

This study is designed as a prospective, controlled, investigator-blinded, parallel-group clinical trial. Fourteen stroke patients aged 18-80 years with hemiplegic shoulder pain will be enrolled and randomized into two groups. After baseline assessment (T0), one group will receive a suprascapular nerve block followed by a standardized physical therapy program, while the control group will receive the same physical therapy program alone. Follow-up assessments will be performed at 2 hours post-intervention (T1, intervention group only), at the end of the 3-week rehabilitation program (T2), and at week 7 (T3).

The primary objective of this study is to evaluate the effect of suprascapular nerve block on shoulder joint proprioception in stroke patients with hemiplegic shoulder pain. Secondary objectives include assessing its effects on pain intensity, shoulder range of motion, post-stroke motor recovery, stroke-specific quality of life, and upper extremity physical function and symptoms.

The null hypothesis is that suprascapular nerve block does not impair shoulder joint proprioception in patients with post-stroke hemiplegic shoulder pain.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* Presence of shoulder pain on the hemiplegic side with a Numeric Rating Scale (NRS) score > 3
* At least 1 month since the cerebrovascular event (subacute and chronic stroke patients)
* Active shoulder flexion range of motion > 90 degrees (required for the application of the laser pointer-assisted joint position sense test)
* First-ever, unilateral hemiplegia

Exclusion Criteria:

* Mini-Mental State Examination score < 24 indicating cognitive impairment
* Presence of aphasia
* Shoulder spasticity with a Modified Ashworth Scale score > 2
* Brunnstrom upper extremity motor stage < 3
* Botulinum toxin type A injection within the last 3 months to muscles affecting shoulder joint movement (trapezius, levator scapulae, pectoralis major, deltoid, serratus anterior, latissimus dorsi, rhomboids, teres major, biceps, coracobrachialis, triceps, supraspinatus, subscapularis, infraspinatus, and teres minor)
* Pre-existing shoulder pathology causing pain in the hemiplegic shoulder
* Presence of neglect syndrome
* Complex regional pain syndrome, central pain, traumatic brachial plexus injury
* Change in pain medication during the study period
* Hypersensitivity to the medication used for suprascapular nerve block (lidocaine)
* Adhesive capsulitis (frozen shoulder)
* Other shoulder pathologies such as fractures or joint replacement

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Laser pointer-assisted joint position sense test | This test will be assessed at baseline (T0). Follow-up assessments will be performed at 2 hours post-intervention (T1, intervention group only), at the end of the 3-week rehabilitation program (T2), and at week 7 (T3)
  The validity and reliability of the laser pointer-assisted joint position sense test in patients with shoulder instability were established by Amir K. Vafadar et al., with inter-observer and intra-observer correlation coefficients of 0.78 and 0.86, respectively. In this test, a laser pointer is secured to the patient's arm using a Velcro strap positioned 5 cm proximal to the elbow. With eyes open, the patient is asked to raise the hemiplegic arm to 90 degrees. The laser point is marked on millimeter paper fixed 1 meter in front of the shoulder joint. The patient is then asked, with eyes open, to relocate the same point to learn the joint position. Subsequently, with eyes closed, the patient is asked to identify the same point again. This second point is marked, and the distance from the initial point is measured along the x- and y-axes. The angular deviation of the shoulder joint position is calculated using the tangent formula.
Thumb localization test | This test will be assessed at baseline (T0). Follow-up assessments will be performed at 2 hours post-intervention (T1, intervention group only), at the end of the 3-week rehabilitation program (T2), and at week 7 (T3)
  For the assessment of proprioception, the thumb localization test will be performed. The validity and reliability of this test in patients with hemiplegia were established by Otaka et al., with a weighted kappa value of 0.84 for inter-observer measurements, indicating high agreement. With the patient's eyes closed, the patient is asked to locate and grasp the thumb of the affected hand using the fingers of the unaffected hand

SECONDARY OUTCOMES:
Numeric Rating Scale (NRS) | This test will be assessed at baseline (T0). Follow-up assessments will be performed at 2 hours post-intervention (T1, intervention group only), at the end of the 3-week rehabilitation program (T2), and at week 7 (T3)
  A 0-10 numeric rating scale will be used to assess pain severity.
Goniometric measurement | This test will be assessed at baseline (T0). Follow-up assessments will be performed at 2 hours post-intervention (T1, intervention group only), at the end of the 3-week rehabilitation program (T2), and at week 7 (T3)
  Shoulder range of motion will be assessed using a standard goniometer, which provides an objective measurement of joint angles in degrees. The goniometer is aligned with anatomical landmarks of the shoulder, and active or passive movements (flexion, abduction, and rotation) are measured according to standardized positioning.
Goal Attainment Scale (GAS) | This test will be assessed at baseline (T0). Follow-up assessments will be performed at 2 hours post-intervention (T1, intervention group only), at the end of the 3-week rehabilitation program (T2), and at week 7 (T3)
  Goal Attainment Scale (GAS) is a goal-oriented functional outcome measure based on the International Classification of Functioning, Disability and Health (ICF) framework and is used to assess the extent to which individuals achieve predefined goals. It quantifies the success or failure of set goals and can be applied in rehabilitation settings. According to this scale, pain during upper extremity dressing was evaluated as follows: -2 = severe pain, -1 = moderate pain, 0 = mild pain, +1 = pain at the end of movement, and +2 = pain-free movement."
Fugl-Meyer Assessment - Upper Extremity | This test will be assessed at baseline (T0). Follow-up assessments will be performed at 2 hours post-intervention (T1, intervention group only), at the end of the 3-week rehabilitation program (T2), and at week 7 (T3)
  Fugl-Meyer Assessment - Upper Extremity: The Fugl-Meyer Upper Extremity Scale is a standardized measure used to evaluate upper extremity motor function after stroke. It is designed to assess movement impairments and loss of muscle control in the upper extremity following stroke. The scale evaluates a range of functions, including shoulder, elbow, wrist, and hand movements, as well as hand use and functional abilities. Each movement is scored on a 0-2 scale, with a maximum total score of 66 points. This scale is widely used in post-stroke rehabilitation programs to assess treatment effectiveness and to monitor motor recovery over time.
Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) questionnaire | This test will be assessed at baseline (T0). Follow-up assessments will be performed at the end of the 3-week rehabilitation program (T2), and at week 7 (T3)
  Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) questionnaire: The QuickDASH is a functional assessment tool used to evaluate upper extremity disability. It is designed to measure symptoms such as pain, weakness, and movement limitations related to the arm, shoulder, and hand, as well as the impact of these problems on activities of daily living. The questionnaire consists of 11 items, each related to a specific activity or function, and patients respond based on their condition over the preceding 7 days. Scoring is divided into two sections: the disability/symptom section (11 items scored from 1 to 5) and an optional high-performance work/sport or music module (4 items scored from 1 to 5). Higher scores indicate greater disability.
Stroke Impact Scale (SIS) | This test will be assessed at baseline (T0). Follow-up assessments will be performed at the end of the 3-week rehabilitation program (T2), and at week 7 (T3)
  The Stroke Impact Scale is a measure used to assess quality of life and functional performance in activities of daily living after stroke. It evaluates patients' physical, psychological, and social functioning. The scale consists of eight domains: strength, activities of daily living/self-care, mobility, hand function, emotion, memory and thinking, communication, and social participation. Each domain assesses different aspects of post-stroke functioning. The SIS is widely used to evaluate the effects of post-stroke treatment and to monitor changes during the recovery process in patients undergoing rehabilitation programs.
Modified Ashworth Scale | This test will be assessed at baseline (T0). Follow-up assessments will be performed at 2 hours post-intervention (T1, intervention group only), at the end of the 3-week rehabilitation program (T2), and at week 7 (T3)
  Modified Ashworth Scale: Shoulder spasticity will be assessed using the Modified Ashworth Scale. Scoring is defined as follows:
  0 = No increase in muscle tone;
  1 = Slight increase in muscle tone, manifested by a catch and release or minimal resistance at the end of the range of motion;
  1+ = Slight increase in muscle tone, manifested by a catch followed by minimal resistance through less than half of the range of motion; 2 = More marked increase in muscle tone through most of the range of motion, but the affected part is easily moved; 3 = Considerable increase in muscle tone, passive movement is difficult; 4 = Affected part rigid in flexion or extension (contracture).

CONTACTS AND LOCATIONS:
Locations (1):
- Fatih Sultan Mehmet Training and Research Hospital Istanbul, İstanbul, Turkey, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Undecided